CLINICAL TRIAL: NCT00529438
Title: A Phase I Dose-finding and Pharmacokinetic Study of RTA 402 (CDDOMe) Administered Orally for 21 Days of a 28-day Cycle in Patients With Advanced Solid Tumors or Lymphoid Malignancies
Brief Title: RTA 402 in Patients With Advanced Solid Tumors or Lymphoid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-0501
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors; Lymphoid Malignancies
MeSH Terms: interventions — bardoxolone methyl

ARMS (1):
- Bardoxolone methyl capsules (Experimental): Bardoxolone methyl to be taken orally for 21 consecutive days, once a day, in the morning prior to food intake.
  Patients to continue to receive treatment for the first 21 days of each 28-day cycle until they experience intolerable toxicity, show evidence of disease progression, or receive a maximum of 18 cycles (18 months).
  Interventions: Drug: Bardoxolone methyl

INTERVENTIONS:
Drug: Bardoxolone methyl
  Other Names: RTA 402

SUMMARY:
This study assesses the tolerability, safety, efficacy and pharmacokinetics of Bardoxolone methyl (RTA 402) in advanced solid tumors and lymphoid malignancies.

DETAILED DESCRIPTION:
Bardoxolone methyl (RTA 402) is a synthetic triterpenoid that has demonstrated significant in vivo single agent anti-cancer activity. This is an open-label phase I dose-escalation study of Bardoxolone methyl (RTA 402) administered orally for the first 21 days of a 28-day cycle.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological documentation of solid tumor or lymphoid malignancy.
* Advanced or metastatic cancer that is either refractory to or have relapsed after standard-of-care curative or survival-prolonging therapy, or for whom no such therapies exist.
* ECOG performance status of less than or equal to 2
* Adequate liver and renal function as documented by the following laboratory test results within 14 days of starting therapy: total bilirubin ≤ 1.5 mg/dL; AST (SGOT) and ALT(SGPT) ≤ 2.5 ULN or ≤ 5 ULN if liver is involved by tumor; serum creatinine ≤2.0 mg/dL OR creatinine clearance >60 mL/min.
* Adequate bone marrow function as documented by the following laboratory test results within 14 days of starting therapy: platelets greater than 100,000/mm3, absolute granulocyte count greater than 1,500/mm3, hemoglobin greater than or equal to 8.0 g/dl.
* Completion of prior chemotherapy, hormonal therapy, radiation therapy, biological therapy, or other investigational cancer therapy, for at least 4 weeks prior to study entry and must have recovered from all acute side effects (to CTC grade 1 or less) prior to initiation of RTA 402. Patients who were receiving mitomycin C or nitrosoureas must be 6 weeks from the last administration of chemotherapy.
* Agree to practice effective contraception during the entire study period.
* Life expectancy of more than 3 months
* Able and willing to sign the informed consent form.
* Willing and able to self-administer orally and document all doses of RTA 402 ingested.

Exclusion Criteria:

* Active brain metastases or primary CNS malignancies.
* Pregnant or breast feeding
* Clinically significant illnesses including, but not limited to: Uncontrolled diabetes; Active or uncontrolled infection; Acute or chronic liver disease; Confirmed diagnosis of HIV infection; Uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, or uncontrolled cardiac arrhythmia.
* Psychiatric illness that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-04-30 (Actual); Primary Completion 2008-12-01 (Actual); Study Completion 2008-12-01 (Actual)

PRIMARY OUTCOMES:
To determine the dose-limiting toxicity, maximum tolerated dose, and recommended phase II dose of Bardoxolone methyl Capsules | 28 day cycles, with a maximum of 18 cycles (18 months)
To characterize the pharmacokinetics of Bardoxolone methyl in this patient population. | 28 day cycles, with a maximum of 18 cycles (18 months)

SECONDARY OUTCOMES:
To document any preliminary antitumor activity. | 28 day cycles, with a maximum of 18 cycles (18 months)
To determine the in vivo molecular and biological effects. | 28 day cycles, with a maximum of 18 cycles (18 months)
To correlate the biological activity of RTA 402 with drug concentration in plasma and blood cellular elements. | 28 day cycles, with a maximum of 18 cycles (18 months)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Case Western Reserve University, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/